CLINICAL TRIAL: NCT00081432
Title: Functional MRI (fMRI) and Diffusion Tensor Imaging (DTI) in Temporal Lobe Epilepsy
Brief Title: Language and Emotional Function in Patients With Temporal Lobe Epilepsy
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040159; 04-N-0159
Record Dates: First submitted 2004-04-10; First posted 2004-04-12 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-04-27

CONDITIONS: Epilepsy; Temporal Lobe
Keywords: Seizures; Language; Memory; Brain; Imaging; Epilepsy; Temporal Lobe Epilepsy
MeSH Terms: conditions — Epilepsy; Seizures; Language; Epilepsy, Temporal Lobe

SUMMARY:
This study uses functional magnetic resonance imaging (fMRI) and diffusion tensor imaging (DTI) to examine how the brain processes tasks involving language and emotion in normal volunteers and in patients with epilepsy. MRI is a diagnostic and research tool that uses a strong magnetic field and radio waves to obtain images of body organs and tissues. The MRI scanner is a metal cylinder surrounded by a magnetic field. During the test, the subject lies on a table that can slide in and out of the cylinder. DTI involves taking pictures of the brain while the subject is at rest in order to learn about the structure of the brain. Information gained from this study will help scientists evaluate the organization of language and emotional functions in the brain.

Normal volunteers and patients with temporal lobe epilepsy 18 years of age and older who are native English speakers and who will undergo surgery for uncontrolled seizures may be eligible for this study. Candidates are initially screened by telephone, then with physical and neurologic examinations and cognitive testing.

The study has two parts, conducted 6 to 12 months apart. Each part consists of the same sets of tests described below, using fMRI and DTI. In patients with epilepsy, Part 1 is scheduled before surgery and Part 2 after surgery.

* fMRI: Subjects are asked to perform two types of tasks while they undergo fMRI. In one task, they are shown pictures of animals and tools and are asked to name them. In a second task, they are shown pictures that range in content from sexually explicit material, to human injury and surgical slides, to pleasant images of children and wildlife and are asked to decide whether they find the pictures pleasant, neutral, or unpleasant.
* DTI: Subjects relax and remain still in the MRI scanner for about 45 minutes.
* Neuropsychological testing: Subjects may be asked to complete questionnaires, take pen-and-paper or computerized tests, and perform motor tasks.

Participants may be asked to repeat the MRI studies, but not the neuropsychological tests, up to four times to investigate different brain functions or to confirm findings.

DETAILED DESCRIPTION:
OBJECTIVES: Epilepsy surgery is emerging as a potent therapeutic intervention for a large group of patients with uncontrolled temporal lobe epilepsy, particularly when performed early in the course of the illness. Seizure freedom is an important goal of seizure surgery, but post-operative neuropsychological functioning is another equally important outcome measure. Both endpoints require careful pre-operative evaluation of the individual patient and better understanding of the functional neuroanatomy of the temporal lobe. In this study fMRI and DTI will be performed in patients with temporal lobe epilepsy and normal volunteers in an attempt to

1. investigate the role of the anterior temporal cortex in semantic processing,
2. evaluate the role of the amygdala in affective processing,
3. correlate the extent of white matter pathway resection with cognitive outcome after temporal lobectomy.

STUDY POPULATION: We plan to study 30 patients with temporal lobe epilepsy (right-sided, left-sided seizure foci) pre and post temporal lobectomy as well as 30 normal volunteers.

DESIGN: The study will be done in two parts both consisting of identical tasks. For the patient group part 1 will be performed prior to temporal lobectomy and part 2, 6-12 months after temporal lobectomy. For the normal volunteer group parts 1 and 2 will be performed at time interval of 6-12 months.

During part 1 all study subjects will undergo neuropsychological evaluation. FMRI will be performed with two tasks: animal and tool naming (to evaluate semantic processing) and rating of emotionally pleasant or unpleasant pictures (to evaluate affective processing). All subjects will also undergo diffusion tensor imaging (DTI) for the visualization of white matter pathways.

During part 2 of the study all of the above tests will be repeated.

FMRI data will be analyzed within the framework of the general linear model in a program such as AFNI 2.5. Statistical comparisons between activation patterns in scans acquired during part 1 and part 2 within either group (intragroup comparison) will be done by voxel wise paired t-test. In a second analysis all 4 groups will be compared in a mixed model. The DTI data will be correlated with the neuropsychological outcome to asses the contribution of white matter abnormalities pre-operatively or severance of white matter pathways post-operative on neuropsychological functioning.

OUTCOME PARAMETERS: Outcome parameters are changes in the fMRI activation pattern post temporal lobectomy and disruption of anisotropy on the diffusion tensor images.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patient Group:

Temporal lobe epilepsy (right-sided, left-sided foci) with or without lesion on a structural MRI scan.

Native English speaker.

Age 18 years or older.

Signed informed consent.

Volunteer Group:

Native English speaker.

Age 18 years or older.

Signed informed consent.

EXCLUSION CRITERIA:

Patient Group:

Medical or technical contraindications to MRI procedures (e.g. no braces, pacemakers, cochlear devices, surgical clips, etc;

History of mental retardation;

Pregnancy;

Claustrophobia;

Inability to comply with the protocol.

Volunteer Group:

Medical or technical contraindications to MRI procedures (e.g. no braces, pacemakers, cochlear devices, surgical clips, etc.);

History of neurologic or psychiatric disease or a learning or attention disorder or mental retardation.

Pregnancy.

Claustrophobia.

Inability to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-04-09; Study Completion 2010-04-27

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Barnes PD. Imaging of the central nervous system in pediatrics and adolescence. Pediatr Clin North Am. 1992 Aug;39(4):743-76. doi: 10.1016/s0031-3955(16)38374-2. PMID 1635805
- [Background] Basser PJ, Pajevic S, Pierpaoli C, Duda J, Aldroubi A. In vivo fiber tractography using DT-MRI data. Magn Reson Med. 2000 Oct;44(4):625-32. doi: 10.1002/1522-2594(200010)44:43.0.co;2-o. PMID 11025519
- [Background] Basser PJ, Pierpaoli C. A simplified method to measure the diffusion tensor from seven MR images. Magn Reson Med. 1998 Jun;39(6):928-34. doi: 10.1002/mrm.1910390610. PMID 9621916